CLINICAL TRIAL: NCT00634738
Title: Neuropathy Along the Median Nerve: Etiology of Symptoms Associated With the Carpal Tunnel Syndrome, a Preliminary Study
Brief Title: The Treatment of the Median Nerve for the Elimination of the Symptoms Associated With the Carpal Tunnel Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guy Hains Chiropractor (Other)
Responsible Party: Guy Hains, UQTR
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: cer-06-115-06.03; no grants
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2010-06

CONDITIONS: Compression Neuropathy, Carpal Tunnel
Keywords: ischemic compression;carpal tunnel syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- one (Experimental)
  Interventions: Procedure: Ischemic Compression (thumb Pressure)

INTERVENTIONS:
Procedure: Ischemic Compression (thumb Pressure) — Pressure, one thumb on the other, applied on the trigger points
  Other Names: Pressure point therapy

SUMMARY:
In carpal tunnel syndrome,trigger points are often found in the biceps muscle,in the aponeurosis of the biceps and in the pronator teres muscle.

We hypothesise that by eliminating these trigger points,using ischemic compressions, may diminish the symptoms.

DETAILED DESCRIPTION:
Using one thumb on the other,the pressure is applied 10 seconds on each TrPs.The treatment is done on each visit for a total of 15(without Charge).

ELIGIBILITY:
Inclusion Criteria:

* Between 20 and 60 years old,
* Numbness in the hand affecting the thumb, the index finger, the middle finger and half the ring finger,
* To have suffered from discomfort on a daily basis for at least three months and to agree to a course of 15 chiropractic treatments at no cost.

Exclusion Criteria:

* History of upper limb or neck surgery,
* Pregnancy and systemic pathologies possibly related to CTS, such as hypothyroidism, diabetes and rheumatoid arthritis.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-01; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Levine DW Questionnaire (J.Bone Joint Surg Am 1993;75:1585-92)on carpal tunnel syndrome | after 15treatments,30 days after,6 months later

SECONDARY OUTCOMES:
A numerical scale,filled by the patient,where they give their perceived improvement from 0% to 100%. | After 15 treatments, 30 days later and 6 months later.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Descarreaux, DC PHD, Study Chair — UQTR
Locations (1):
- Guy Hains 2930 Côte RIchelieu, Trois-Rivières, Quebec, Canada